CLINICAL TRIAL: NCT06371807
Title: Immunogenicity Profile of Neoadjuvant Keytruda in Combination With Anthracycline Versus Carboplatin/PAclitaxel Containing Chemotherapy Regimen for The Treatment of Early-stage, TILs-Positive, Triple-Negative Breast CanceR
Brief Title: Trial for Treatment of High Risk BC With Two Sequences of Neoadjuvant Chemotherapy With Pembrolizumab
Acronym: KEYPARTNER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacao Champalimaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU CTR n.º 2023-507008-30-00
Record Dates: First submitted 2024-03-12; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-02

CONDITIONS: Early Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — pembrolizumab; Doxorubicin; Epirubicin; Cyclophosphamide; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: (KXCb - PA[E]C) (Active Comparator): Pembrolizumab (K) every 3 weeks (Q3W) + paclitaxel (X) + carboplatin (Cb) once weekly (QW) for 4 cycles in the neoadjuvant setting followed by pembrolizumab + doxorubicin or epirubicin (A or E) + cyclophosphamide (C) for 4 cycles followed by pembrolizumab every 6 weeks for 5 cycles (total of 1 year of pembrolizumab) in the adjuvant setting.
  Interventions: Drug: Pembrolizumab injection
- (KPA[E]C - KXCb) (Experimental): Pembrolizumab + doxorubicin or epirubicin (A or E) + cyclophosphamide (C) for 4 cycles in the neoadjuvant setting followed by pembrolizumab (K) every 3 weeks (Q3W) + paclitaxel (X) + carboplatin (Cb) once weekly (QW) for 4 cycles followed by pembrolizumab every 6 weeks for 5 cycles (total of 1 year of pembrolizumab) in the adjuvant setting
  Interventions: Drug: Pembrolizumab injection

INTERVENTIONS:
Drug: Pembrolizumab injection — (KXCb - PA[E]C) vs (KPA[E]C - KXCb) Pembrolizumab (K) + paclitaxel (X) + carboplatin (Cb) followed by pembrolizumab + doxorubicin or epirubicin (A or E) + cyclophosphamide (C) followed by pembrolizumab in the adjuvant setting vs Pembrolizumab + doxorubicin or epirubicin (A or E) + cyclophosphamide (C) followed by pembrolizumab (K) + paclitaxel (X) + carboplatin (Cb) followed by pembrolizumab in the adjuvant setting
  Other Names: Doxorubicin or Epirubicin; Cyclophosphamide; Paclitaxel; Carboplatin

SUMMARY:
Phase II, randomized, Active-controlled open label trial for treatment of high risk, HR-/HER2- (triple negative) breast cancer, with two sequences of neoadjuvant chemotherapy on a background of pembrolizumab

DETAILED DESCRIPTION:
This is a randomized, open-label, pilot study to evaluate the existence of a differential tumor immunomodulatory profile of neoadjuvant pembrolizumab in combination with paclitaxel and carboplatin vs pembrolizumab in combination with EC/AC in patients with triple negative, tumor infiltrating lymphocytes (TILs) enriched, early breast cancer to allow the optimization of future de-escalation strategies. There will be crossover between treatment arms when moving from the neoadjuvant to adjuvant treatment period for completion of standard chemotherapy plus pembrolizumab.

The chemotherapy regimen included in this study is built upon previous studies of pembrolizumab plus chemotherapy. The synergistic effect of different chemotherapy backbone and pembrolizumab will be studied as part of a 2-arm study:

Arm 1: (KXCb - PA[E]C): Pembrolizumab (K) every 3 weeks (Q3W) + paclitaxel (X) + carboplatin (Cb) once weekly (QW) for 4 cycles in the neoadjuvant setting followed by pembrolizumab + doxorubicin or epirubicin (A or E) + cyclophosphamide (C) for 4 cycles followed by pembrolizumab every 6 weeks for 5 cycles (total of 1 year of pembrolizumab) in the adjuvant setting.

Arm 2: (KPA[E]C - KXCb): Pembrolizumab + doxorubicin or epirubicin (A or E) + cyclophosphamide (C) for 4 cycles in the neoadjuvant setting followed by pembrolizumab (K) every 3 weeks (Q3W) + paclitaxel (X) + carboplatin (Cb) once weekly (QW) for 4 cycles followed by pembrolizumab every 6 weeks for 5 cycles (total of 1 year of pembrolizumab) in the adjuvant setting.

In case of clinical evidence of non-pCR, i.e., biopsy proven residual disease after the neoadjuvant phase, patients can proceed to the crossover part of the adjuvant phase before surgery (i.e., 4 cycles of chemotherapy plus pembrolizumab) receiving the remaining administrations of pembrolizumab after surgery.

ELIGIBILITY:
Inclusion Criteria: Participants are eligible to be included in the study only if all the following criteria apply:

1. Be willing and able to provide written informed consent for the trial. The subject may also provide consent for Future Biomedical Research. However, the subject may participate in the main trial without participating in Future Biomedical Research.
2. Be a female or male participant who is at least 18 years of age on the day of signing informed consent.
3. Have locally histologically confirmed diagnosis of invasive carcinoma of the breast that is classified as TNBC, as defined by the most recent ASCO/CAP guidelines.
4. Has locally confirmed tumor infiltrating lymphocytes (stromal) (sTILs) equal to or above 10%, as defined by the most recent International Guidelines on TIL Assessment in Breast Cancer.
5. Have previously untreated non-metastatic (M0) TNBC defined as the following combined primary tumor (T) and regional lymph node (N) staging per current AJCC staging criteria for breast cancer staging criteria as assessed by the investigator based on radiological and/or clinical assessment:

   1. T1c, N1-N2
   2. T2, N0-N2
   3. T3, N0-N2
   4. T4a-d, N0-N2 Note: bilateral tumors (ie, synchronous cancers in both breasts) and/or multi-focal (ie, 2, separate lesions in the same quadrant)/multi-centric (ie, 2 separate lesions in different quadrants) tumors are allowed, as well as inflammatory breast cancer, and the tumor with the most advanced T stage should be used to assess the eligibility. If the subject has either bilateral or multi-focal/multi-centric disease, TNBC needs to be confirmed in at least 2 lesions/breast/focus. Beyond this rule, the extent of tumor biopsy confirmation is based on the best clinical judgment by local investigators.
6. Provide a core needle biopsy consisting of at least 3 separate tumor cores from the primary tumor at screening to the designated central biobank (or responsible laboratories) and is willing to provide a second biopsy at the end of the first cycle of treatment.

   Note: Detailed instructions on sample collection, processing, storage and shipment to the central biobank are provided in the Laboratory Manual.
7. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 performed within 10 days of treatment initiation.
8. Have left ventricular ejection fraction (LVEF) of ≥50% or ≥ institution lower limit of normal (LLN) as assessed by echocardiogram (ECHO) or multigated acquisition (MUGA) scan performed at screening.
9. Have adequate organ function as defined in the following table (Table 2). Specimens must be collected within 28 days prior to the start of study intervention.
10. Male participants:

A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 12 months after the last dose of cyclophosphamide or 6 months after last chemotherapy (whichever occurs last) and refrain from donating sperm during this period.

Female participants:

A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

a. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR b. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 12 months after the last dose of cyclophosphamide or 6 months after last chemotherapy (whichever occurs last).

-

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
2. Has received prior chemotherapy, targeted therapy, and radiation therapy within the past 12 months.
3. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
4. Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 4 weeks of the first dose of treatment in this current trial.

   Note: subject should be excluded if he/she received an investigational agent with anticancer or anti-proliferative intent within the last 12 months.
5. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
7. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
8. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
9. Has significant cardiovascular disease, such as:

   1. History of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the last 6 months
   2. Congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV or history of CHF NYHA class III or IV
10. Has a known history of Human Immunodeficiency Virus (HIV) infection.
11. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
12. Has a known history of active TB (Bacillus Tuberculosis).
13. Has an active infection requiring systemic therapy.
14. If surgery was performed prior to screening, has persistent adverse events or incomplete wound healing considered clinically relevant by the treating investigator.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through at least 12 months after the last dose of cyclophosphamide or 6 months after last chemotherapy (whichever occurs last).
18. Has had an allogenic tissue/solid organ transplant.
19. Subjects without legal capacity who are unable to understand the nature, scope, significance and consequences of this clinical trial and to consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Detect immunologic activation signal and the immunologically defined most suitable patient population for the synergistic interaction between pembrolizumab and chemotherapy backbone | At the end of cycle 1 (each cycle is 28 days)
  Compare signals of immunological activation or a more favorable immunological context beetween T cell subpopulations and transcriptional changes of T cell populations infiltrating tumors at baseline and C2D1
Rate of pCR | 6 months to one year after subject inclusion
  Compare the rate of pCR in subjects with locally advanced TNBC with TILs ≥ 10% in arm A and arm B at cycle 4
Primary translational endpoint | 6 months to one year after subject inclusion
  Quantification of number of T cells per mm2 with different phenotypes using fate bifurcation as defined as the proportion of TILs with the phenotype T-bet(hi) PD1(mid) CD8+.

SECONDARY OUTCOMES:
Changes in the immunogenic phenotype | 6 months to one year after subject inclusion
  Determine changes in the immunogenic phenotype by longitudinally evaluating RNA-based gene expression signatures (e.g., tumor inflammation signature expression of granzyme A [GZMA] and perforin 1 at baseline and at C2D1.
Incidence of treatment relatred Adverse events | 6 months to one year after subject inclusion
  Describe the safety and tolerability of the combinations of pembrolizumab plus chemotherapy (either EC/AC or paclitaxel + carboplatin) in the Neoadjuvant and Adjuvant setting throught the CTCAE version 5.0 adverse event evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Cardoso, MD, Study Director — Breast Unit Director
Locations (3):
- Portugal (3):
  - Fundaçao Champalimaud, Avenida Brasilia,, Lisbon
  - Centro Hospitalar Universitário Lisboa Norte E.P.E, Lisbon
  - Instituto Português de Oncologia Francisco Gentil, E.P.E, Porto

IPD SHARING:
Plan to Share IPD: Yes
Primary outcome will be shared in major medical Congress
Supporting Information: Study Protocol, SAP
Time Frame: Within one year of primary analysies